CLINICAL TRIAL: NCT03280472
Title: Transition to College/Miami University
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Miami University (Other)
Responsible Party: Principal Investigator, Elise Clerkin, Assistant Professor, Miami University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01368r
Record Dates: First submitted 2017-08-30; First posted 2017-09-12 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Interpretation Bias Modification; Symptom Tracking
Keywords: Interpretation Bias; Interpretation Modification Program

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Bias Modification (Experimental): Participants will complete three session of cognitive bias modification.
  Interventions: Behavioral: Cognitive Bias Modification
- Symptom Tracking (Other): Participants will track their symptoms.
  Interventions: Behavioral: Symptom tracking

INTERVENTIONS:
Behavioral: Cognitive Bias Modification — CBM training. For those in the CBM condition, participants will complete a task. In this task, they will read ambiguous, two- to four-sentence social-related scenarios on the computer. The final word in the scenario will have a missing letter. Participants will type the missing letter. Participants will also be asked to answer a "Yes/No" comprehension question about the scenario. The missing letter will "resolve" the ambiguity of the scenario in a positive way, intended to train participants to have more positively-biased interpretations of ambiguous social information
  Arms: Cognitive Bias Modification
Behavioral: Symptom tracking — Participants will track their symptoms
  Arms: Symptom Tracking

SUMMARY:
The current project will test whether a computerized training program, Cognitive Bias Modification (CBM), can be used as a prevention inoculation tool to reduce vulnerability to anxiety among incoming college students. Those not in the CBM condition will complete a symptom tracking condition (ST). We will also test whether ST influences vulnerability to anxiety among incoming college students.

ELIGIBILITY:
Inclusion Criteria:

* First and Second year students
* Entered college in fall of 2017
* Fluent in English
* LSAS-SR score greater than or equal to 14 and less than or equal to 74.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-09-18 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Change in Student Adjustment to College Questionnaire | Participants report on their past few days. The SACQ is administered at T1-T5. T2 occurs within ~1 week of T1/baseline. T2-T5 are spaced ~1 week apart from each other. Sessions are ~60-90 minutes.
  Self-report on the degree to which the participant feels they are transitioning to college successfully.

SECONDARY OUTCOMES:
Change in Interpretations | Participants report interpretations to a variety of situations. The IQ is administered at T1 and T4. T2 occurs within 1 week of T1/baseline. T2-T5 are spaced ~1 week apart from each other. Sessions are ~60-90 minutes.
  A questionnaire assessing their interpretation of ambiguous, potentially anxiety-provoking situation
Change in Liebowitz Social Anxiety Scale-Self-Report | Participants report on symptoms during the past week. The LSAS-SR is administered at T1-T5. T2 occurs within ~1 week of T1/baseline. T2-T5 are spaced ~1 week apart from each other. Sessions are ~60-90 minutes.
  Self-report of social anxiety symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Elise Clerkin, PhD, Principal Investigator — Miami University
Locations (1):
- Anxiety Cognition and Emotion Laboratory, Oxford, Ohio, United States

IPD SHARING:
Plan to Share IPD: No